CLINICAL TRIAL: NCT00210678
Title: An Observational Study to Evaluate Intravaginal Ejaculatory Latency Time and Patient-Reported Outcomes in Men With and Without Premature Ejaculation
Brief Title: A Study to Evaluate Intravaginal Ejaculation Time in Men With and Without Premature Ejaculation
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004225; R096769-PRE-3004 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Dapoxetine; Premature ejaculation; Ejaculation; Sexual dysfunction; Orgasmic disorder
MeSH Terms: conditions — Erectile Dysfunction; Premature Ejaculation; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group: 1: Men with premature ejaculation (PE)
  Interventions: Behavioral: No intervention
- Group: 2: Men without PE
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: No intervention — No treatment is given to the patients as this is an observational study.

SUMMARY:
The purpose of the study is to characterize intravaginal ejaculatory latency time (time between the start of vaginal intercourse and the start of intravaginal ejaculation) in men with and without premature ejaculation (PE) and to assess the validity of patient-reported outcomes.

DETAILED DESCRIPTION:
This is a multinational, multicenter, observational study in men with and without PE. The study consists of three visits: one visit for screening and enrollment, and two visits for observation after 1 and 2 months (total duration of 8 weeks). No study treatment for PE is administered to patients during the course of the study. Patients and their partners are expected to attempt sexual intercourse at least 2 times a week during the 8-week study period and to use a stopwatch to record the intravaginal ejaculatory latency time (IELT) during intercourse. At visits during the observation period "patients" (and/or partners if partners are responsible for completing questionaires) also provide patient-reported outcomes (PROs) by answering several questionnaires that include the topics of control over ejaculation, satisfaction with sexual intercourse, personal distress, interpersonal difficulty, and self-esteem. The study will estimate the distribution of the average IELT values for men with PE and men without PE.

ELIGIBILITY:
Inclusion Criteria:

* Must be in a stable, monogamous, sexual relationship with the same woman (18 years of age or older) for at least 6 months, who plan to maintain their relationship for the duration of the study
* Must be in good general health
* Patient and partner willing to avoid situations or activities that may have an effect on their sexual activity (eg, refrain from any preplanned surgery)

Exclusion Criteria:

* Has history of drug abuse within the past 2 years
* Has history of or current major psychiatric disorder such as mood disorders, anxiety disorders, schizophrenia, other psychotic disorders, or alcoholism
* Must have erectile dysfunction
* Patient who has decreased interest in sexual intercourse or has other forms of sexual dysfunction
* Patient whose partner has decreased interest in sexual intercourse, painful intercourse, or other forms of female sexual dysfunction
* Patient whose partner is more than 3 months pregnant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One thousand patients (at least 200 men with premature ejaculation (PE) and at least 800 men without PE) will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1115 (Actual)
Dates: Start 2005-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change in Intravaginal Ejaculatory Latency Time (IELT) | Day 1 to Week 8
  Estimated distribution of the average IELT for both the premature ejaculation (PE) and non-PE populations will be calculated.
Change in Patient-Reported Outcomes (PRO) | Week 4 and Week 8
  Additional evidence of reliability and validity of PROs for patients with and without PE and their partners will be expolred. The PROs will include different parameters related to (control over ejaculation, satisfaction with sexual intercourse, personal distress, and interpersonal difficulty).

SECONDARY OUTCOMES:
Association between intravaginal ejaculatory latency time (IELT) and patient reportedout comes (PROs) | Up to Week 8
  Association between IELT and PROs used in this study will be explored.
Utility of the Male Sexual Function Scale and Ejaculation Questionnaires | Day 1
  The study will explore utility of the Male Sexual Function Scale and Ejaculation Questionnaire as screening instruments.
PROs and IELT as indicators to clasify PE status. | Up to Week 8
  The study will evaluate the ability of PROs and IELT to classify PE status

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.